CLINICAL TRIAL: NCT06588491
Title: KYSA-8: A Phase 2 Open-Label, Single-Arm, Multicenter Study of KYV-101, an Autologous Fully Human Anti-CD19 Chimeric Antigen Receptor T-Cell (CD19 CAR T) Therapy, in Subjects With Treatment Refractory Stiff Person Syndrome
Brief Title: KYSA-8: A Study of Anti-CD19 Chimeric Antigen Receptor T-Cell (CD19 CAR T) Therapy, in Subjects With Treatment Refractory Stiff Person Syndrome
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Kyverna Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KYSA-8; KYV101-008 (Other: Kyverna Therapeutics)
Record Dates: First submitted 2024-09-06; First posted 2024-09-19 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Stiff-Person Syndrome; SPS
Keywords: SPS; Stiff-Person Syndrome
MeSH Terms: conditions — Stiff-Person Syndrome | interventions — Cyclophosphamide; fludarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- KYV-101 CAR-T cells with lymphodepletion conditioning (Experimental): Dosing with KYV-101 CAR T cells
  Interventions: Biological: Standard lymphodepletion regimen

INTERVENTIONS:
Biological: Standard lymphodepletion regimen — Standard lymphodepletion regimen
  Other Names: Cyclophosphamide; Fludarabine

SUMMARY:
A Study of Anti-CD19 Chimeric Antigen Receptor T-Cell Therapy for Subjects with Treatment Refractory Stiff Person Syndrome

DETAILED DESCRIPTION:
Stiff person syndrome (SPS) is a rare progressive immune-mediated disorder of the central nervous system (CNS) that is characterized by progressive rigidity and painful spasms of predominantly axial and proximal limb muscles. The condition gradually worsens over time and left untreated, it can lead to permanent disability and in some cases, mortality.

B cells contribute to systemic autoimmunity and development of disease in several ways, most notably via cytokine production, antigen presentation and complement activation (via autoantibody production). In SPS, B cell involvement is supported by the presence of antibodies against glutamic acid decarboxylase (GAD), which is widely expressed within the CNS, catalyzing the conversion of the excitatory neurotransmitter l-glutamate to the inhibitory GABA.

CAR-T therapy such as KYV-101 may be an effective treatment for SPS, by targeting these autoreactive B cells. Using chimeric antigen receptor (CAR) T-cell technology, engineered T cells with receptors are designed to recognize and eliminate B cells, including those that produce GAD autoantibodies. This approach aims to intervene at the root of the autoimmune response, offering a precise and potentially transformative treatment for SPS. CAR-T cell therapy holds promise as a targeted and effective intervention, addressing the autoimmune component directly and potentially halting disease progression.

ELIGIBILITY:
Key Inclusion Criteria:

* Subject must have been diagnosed SPS per the following criteria:

  * Rigidity of limb and axial (trunk) muscles prominent in the abdominal and thoracolumbar paraspinal areas and making bending difficult
  * Clinical or electrophysiological evidence of continuous contraction of agonist and antagonist muscles
  * Episodic spasms precipitated by unexpected noises, tactile stimuli, or emotional upset
  * Absence of any other neurologic disease that could explain the stiffness and rigidity
  * High titer serum anti-GAD65 antibodies shown at screening -OR- seropositive for anti-glycine antibodies. If anti-GAD65 antibodies are lower than the high titer threshold peripherally but positive in the cerebrospinal fluid (CSF), the subject can be included. A prior documented high titer anti-GAD65 antibody level may be acceptable subject to sponsor review.
* Active symptoms with inadequate response to at least one immunomodulatory therapy.
* Stiffness index ≥2.
* At least 20 of the 25 enrolled subjects should be ambulatory.

Key Exclusion Criteria:

* Bedridden subjects for more than 3 months.
* History of CNS or spinal cord tumor, metabolic or infectious cause of myelopathy, genetically inherited progressive CNS disorder, sarcoidosis, non-SPS progressive neurologic condition or progressive multifocal leukoencephalopathy (PML).
* History of stroke, seizure, dementia, Parkinson's disease, cerebellar diseases, psychosis, aphasia, and any other neurologic disorder that is of a nature and severity that the investigator considers would increase the risk for the subject.
* Cardiac ejection fraction ≤ 40%.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2024-09-25 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
To evaluate efficacy of KYV-101 | Up to 12 months
  Change in the Timed 25-Foot Walk (T25-FW) from baseline
To evaluate the safety of KYV-101 | Up to 12 months
  Incidence of adverse events and laboratory abnormalities

SECONDARY OUTCOMES:
To evaluate efficacy of KYV-101 | Up to 12 months
  Change in Modified Rankin Scale from baseline Modified Rankin Scale: Scoring is from 0 (no symptoms) to 6 (death). A higher score indicates a worse outcome.
To evaluate efficacy of KYV-101 | Up to 12 months
  Change in the scores of the distribution-of-stiffness index from baseline. Distribution of Stiffness Index: Scoring is from 0 to 6. A higher score indicates a worse outcome.
To evaluate efficacy of KYV-101 | Up to 12 months
  Change in Hauser Ambulation Index. Hauser Ambulation Index: Scoring is from 0 to 9. A higher score indicates a worse outcome.
To evaluate efficacy of KYV-101 | Up to 12 months
  Change in Heightened sensitivity scale. Heightened Sensitivity Scale: Scoring is from 0 to 7. A higher score indicates a worse outcome.

OTHER OUTCOMES:
To evaluate efficacy of KYV-101 | Up to 12 months
  6-minute walk test
To evaluate efficacy of KYV-101 | Up to 12 months
  Change in anti-GAD-65 antibody levels
To evaluate efficacy of KYV-101 | Up to 12 months
  Change in anti-glycine receptor antibodies
To evaluate efficacy of KYV-101 | Up to 12 months
  36-Short form survey (SF-36). The SF-36 has eight scaled scores. Scores range from 0 - 100 with lower scores equating to more disability and higher scores equating to less disability.
To characterize the pharmacokinetics (PK) | Up to 12 months
  Levels of KYV-101 CAR-positive T cells in the blood
To evaluate the immunogenicity (humoral response) of KYV-101 | Up to 12 months
  Percentage of participants who develop anti-KYV-101 antibodies by immunoassays
To characterize the pharmacodynamics (PD) | Up to 12 months
  Levels of systemic cytokine concentrations in serum
To characterize the pharmacodynamics (PD) | Up to 12 months
  Levels of B cells in the blood

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Kyverna Therapeutics
Locations (3):
- United States (3):
  - University of Colorado Anschutz Medical Campus, Aurora, Colorado
  - Mayo Clinic, Rochester, Minnesota
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dalakas MC. Therapies in Stiff-Person Syndrome: Advances and Future Prospects Based on Disease Pathophysiology. Neurol Neuroimmunol Neuroinflamm. 2023 Apr 14;10(3):e200109. doi: 10.1212/NXI.0000000000200109. Print 2023 May. PMID 37059468
- [Background] Duddy ME, Baker MR. Stiff person syndrome. Front Neurol Neurosci. 2009;26:147-165. doi: 10.1159/000212375. Epub 2009 Apr 6. PMID 19349711